CLINICAL TRIAL: NCT05037630
Title: Feasibility Evaluation of a Self-guided Digital Tool for Problematic Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Martin Kraepelien, Licensed clinical psychologist, Principal investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCOHOLDIARY1
Record Dates: First submitted 2021-08-27; First posted 2021-09-08 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-guided Digital Tool for Problematic Alcohol Use (Experimental): Self-guided Digital Tool for Problematic Alcohol Use during 8 weeks with clinical telephone interviews pre ant post intervention.
  Interventions: Behavioral: Self-guided Digital Tool for Problematic Alcohol Use

INTERVENTIONS:
Behavioral: Self-guided Digital Tool for Problematic Alcohol Use — See arm/group-description
  Other Names: ALVA

SUMMARY:
The purpose of the study is to evaluate the feasibility of a new monitored self-guided digital intervention based on an alcohol diary and techniques from cognitive behavioral therapy and relapse prevention. The participants will be adults with problematic alcohol use. An uncontrolled trial will explore participant's usability and treatment credibility ratings, behavioural engagement and preliminary effects on alcohol use.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Access to internet
3. ≥8 points for men and ≥6 points for women on Alcohol Use Disorders Identification Test (AUDIT)

Exclusion Criteria:

1. Insufficient knowledge of the Swedish language
2. Difficulties reading or writing related to a digital intervention.
3. Other ongoing psychological treatment with a content similar to that in the current study (problematic alcohol use).
4. High suicide risk based on telephone assessment.
5. Other urgent need for more intensive psychiatric care, or addiction care services, based on telephone assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Standardized drinks per week (based on Time Line Follow Back) | 3 months after intervention
  Changes in standardized drinks per week (using Time Line Follow Back)
Heavy drinking days (based on Time Line Follow Back) | 3 months after intervention
  Changes in number of heavy drinking days (defined as ≥ 5 (men) or ≥ 4 (women) standardized drinks on a single day, using the Time Line Follow Back)

SECONDARY OUTCOMES:
Standardized drinks per week (based on Time Line Follow Back) | Immediately after the intervention
  Changes in standardized drinks per week (using Time Line Follow Back)
Heavy drinking days (based on Time Line Follow Back) | Immediately after the intervention
  Changes in number of heavy drinking days (defined as ≥ 5 (men) or ≥ 4 (women) standardized drinks on a single day, using the Time Line Follow Back)
Diagnostic criteria Alcohol Use Disorder | 3 months after intervention
  Using SCID-5
Diagnostic criteria Alcohol Use Disorder | Immediately after the intervention
  Using SCID-5
System Usability Scale | Immediately after the intervention
  System Usability Scale (SUS), score range 0-100, higher is better.
Credibility/Expectancy questionnaire | Immediately after the intervention
  Credibility/Expectancy questionnaire, score range 0-50, higher is better
Alcohol Use Disorders Identification Test | 3 months after intervention
  Alcohol Use Disorders Identification Test (AUDIT), score range 0-40, lower is better
Alcohol Use Disorders Identification Test | Immediately after the intervention
  Alcohol Use Disorders Identification Test (AUDIT), score range 0-40, lower is better
Brunnsviken Brief Quality of Life Scale | 3 months after intervention
  Brunnsviken Brief Quality of Life Scale (BBQ), score range 0-96, higher is better
Brunnsviken Brief Quality of Life Scale | Immediately after the intervention
  Brunnsviken Brief Quality of Life Scale (BBQ), score range 0-96, higher is better
Penn Alcohol Craving Scale | 3 months after intervention
  Penn Alcohol Craving Scale (PACS), score range 0-30, lower is better
Penn Alcohol Craving Scale | Immediately after the intervention
  Penn Alcohol Craving Scale (PACS), score range 0-30, lower is better
Patient Health Questionnaire 9 | 3 months after intervention
  Patient Health Questionnaire 9 (PHQ-9), score range 0-27, lower is better
Patient Health Questionnaire 9 | Immediately after the intervention
  Patient Health Questionnaire 9 (PHQ-9), score range 0-27, lower is better
Generalized Anxiety Disorder 7 | 3 months after intervention
  Generalized Anxiety Disorder 7 (GAD-7), score range 0-21, lower is better
Generalized Anxiety Disorder 7 | Immediately after the intervention
  Generalized Anxiety Disorder 7 (GAD-7), score range 0-21, lower is better

OTHER OUTCOMES:
Behavioral engagement | Immediately after the intervention
  Number of alcohol diary entries
Telephone interview on perceptions of intervention | Immediately after the intervention
  Quotes

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum för Psykiatriforskning, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraepelien M, Sundstrom C, Johansson M, Ivanova E. Digital psychological self-care for problematic alcohol use: feasibility of a new clinical concept. BJPsych Open. 2023 May 24;9(3):e91. doi: 10.1192/bjo.2023.73. PMID 37222099